CLINICAL TRIAL: NCT03955952
Title: Cardiovascular Outcomes in Patients With Type 2 Diabetes and Obesity: Comparison of Metabolic Surgery Versus Usual Care
Brief Title: Cardiovascular Outcomes in Bariatric Surgery Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ali Aminian, Principal Investigator, The Cleveland Clinic
Other Study IDs: 19-066
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Obesity; Type2 Diabetes; Bariatric Surgery Candidate
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric Surgery: Patients with type 2 diabetes with BMI >=30 that underwent bariatric surgery
  Interventions: Procedure: Bariatric Surgery
- Non-Surgical Control: Matched non-surgical controls with type 2 diabetes and BMI >=30

INTERVENTIONS:
Procedure: Bariatric Surgery — Patients chosen using the following codes:
  Current Procedural Terminology (CPT): 43633, 43634, 43770, 43775, 43644, 43645, 43659, 43842, 43843, 43844, 43845, 43846, 43847 International Classification of Diseases (ICD): 44.31, 43.82,44.95, 43.89, 44.38, 44.39, 44.68 Healthcare Common Procedure Coding System (HCPCS): S2082, S2085
  Groups: Bariatric Surgery

SUMMARY:
The objective of the analysis was to evaluate the relationship between bariatric surgery and cardiovascular outcomes in obese patients with type 2 diabetes. This is a retrospective matched cohort study of patients with diabetes that underwent bariatric surgery at the Cleveland Clinic between 2004-2017. Each bariatric patient was matched to a non-surgical control with obesity and type 2 diabetes in a 1:5 ratio using data from the Electronic Medical Record (EMR). The maximum observation time was 10 years. Cumulative incidence rates for all-cause mortality and cardiovascular events were calculated at years 1, 3, 5, 7 and 10. Kaplan-Meier curves were created for all the outcomes with all-cause mortality considered as a completing risk.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes
* 18-80 years old
* BMI>=30
* HBA1c >6.4 OR taking at lease one (1) diabetes medication (insulin or non-insulin)

Exclusion Criteria:

* History of liver, heart, or lung transplant
* Emergency department admission within 5 days prior
* Cancer diagnosis within 1 year prior
* Any prior ejection fraction <20%
* Non-surgical controls were excluded if they died within 30 days after the index date (date of surgery for the bariatric patients)
* Last follow-up date on or before the index date

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes patients with obesity (BMI>=30) between 18-80 years old.
Sampling Method: Probability Sample
Enrollment: 13722 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Composite of All-Cause Mortality and Cardiovascular Outcomes | From index date through a maximum of 10 years
  Time to first occurrence of all-cause mortality, coronary artery disease event, stroke, heart failure, nephropathy, or atrial fibrillation

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Event (MACE-3) | From index date through a maximum of 10 years
  Time to first occurrence of all-cause mortality, myocardial infarction or ischemic stroke
All-Cause Mortality | From index date through a maximum of 10 years
  Time to occurrence of death from any cause
Incidence of Coronary Disease Events | From index date through a maximum of 10 years
  Time to first occurrence of myocardial infarction, unstable angina, percutaneous coronary intervention, or coronary artery bypass grafting
Incidence of Cerebrovascular Events | From index date through a maximum of 10 years
  Time to first occurrence of ischemic or hemorrhagic stroke, carotid stenting or endarterectomy
Incidence of Heart Failure | From index date through a maximum of 10 years
  Time to first occurrence of heart failure
Development of Nephropathy | From index date through a maximum of 10 years
  Time to first occurrence of nephropathy defined as >=2 measures of estimated Glomerular Filtration Rate (eGFR) <60 ml/min/1.73m^2 separated by at least 90 days without intervening values >=60
Incidence of Atrial Fibrillation | From index date through a maximum of 10 years
  Time to first occurrence of atrial fibrillation defined by the following codes:
  International Classification of Diseases ICD-9: 427.31 ICD-10: i48.0, i48.1, i48.2, i48.91 Current Procedural Terminology (CPT): 93650, 93653, 93656, 93657

OTHER OUTCOMES:
Percentage Change in Body Weight | 1,3 and 5 years post-index date
  Percentage change in body weight from index date to years 1, 3 and 5 post-index date
Percentage Change in Hemoglobin A1c | 1,3 and 5 years post-index date
  Percentage change in hemoglobin A1c from index date to years 1, 3 and 5 post-index date
Percentage Change in Systolic Blood Pressure (SBP) | 1,3 and 5 years post-index date
  Percentage change in SBP from index date to years 1, 3 and 5 post-index date
Percentage Change in Diastolic Blood Pressure (DBP) | 1,3 and 5 years post-index date
  Percentage change in DBP from index date to years 1, 3 and 5 post-index date
Percentage Change in High Density Lipoprotein (HDL) | 1,3 and 5 years post-index date
  Percentage change in HDL from index date to years 1, 3 and 5 post-index date
Percentage Change in Low Density Lipoprotein (LDL) | 1,3 and 5 years post-index date
  Percentage change in LDL from index date to years 1, 3 and 5 post-index date
Percentage Change in Triglycerides | 1,3 and 5 years post-index date
  Percentage change in triglycerides from index date to years 1, 3 and 5 post-index date

CONTACTS AND LOCATIONS:
Overall Officials: Phil Schauer, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aminian A, Zajichek A, Arterburn DE, Wolski KE, Brethauer SA, Schauer PR, Kattan MW, Nissen SE. Association of Metabolic Surgery With Major Adverse Cardiovascular Outcomes in Patients With Type 2 Diabetes and Obesity. JAMA. 2019 Oct 1;322(13):1271-1282. doi: 10.1001/jama.2019.14231. PMID 31475297